CLINICAL TRIAL: NCT02890693
Title: Improving Cardio-metabolic and Mental Health in Women With Gestational Diabetes Mellitus (GDM) and Their Offspring: MySweetHeart Trial
Brief Title: Improving Cardio-metabolic and Mental Health in Women With Gestational Diabetes Mellitus and Their Offspring
Acronym: MySweetHeart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Jardena Puder, Professor, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-00745
Record Dates: First submitted 2016-08-05; First posted 2016-09-07 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Gestational Diabetes Mellitus
Keywords: gestational diabetes mellitus; randomized controlled trial; lifestyle intervention; cardiovascular; metabolic; mental health; depression; physical activity; dietary intervention
MeSH Terms: conditions — Diabetes, Gestational; Psychological Well-Being; Depression; Motor Activity | interventions — Psychosocial Intervention; Exercise; Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- interdisciplinary lifestyle/psychosocial (Experimental): The multidimensional interdisciplinary lifestyle and psychosocial intervention will be offered on top of usual care. It will consist of individual sessions (face-to-face or telephone contact) with different members of the interdisciplinary team (dietician, physiotherapist, clinical psychologist or coach) and two group sessions.
  Interventions: Behavioral: interdisciplinary lifestyle and psychosocial intervention
- treatment as usual (No Intervention): Usual clinical follow-up and treatment is based on the current American Diabetes Association, the Endocrine Society guidelines, and the NICE guidelines.

INTERVENTIONS:
Behavioral: interdisciplinary lifestyle and psychosocial intervention — The multidimensional interdisciplinary lifestyle and psychosocial intervention will be offered on top of usual care. It will consist of individual sessions (face-to-face or telephone contact) with different members of the interdisciplinary team (dietician, physiotherapist, clinical psychologist or coach) and two group sessions. It will take place during pregnancy and during the first year postpartum.
  Other Names: lifestyle intervention; physical activity; dietary intervention; psychosocial intervention
  Arms: interdisciplinary lifestyle/psychosocial

SUMMARY:
MySweetHeart Trial is a randomized controlled trial to test the effect of a multidimensional interdisciplinary lifestyle and psychosocial intervention to improve the cardio-metabolic and mental health of women with GDM and their offspring.

Primary objective of MySweetHeart Trial:

To test the effect of a multidimensional interdisciplinary lifestyle and psychosocial intervention in women with GDM to improve 1) their metabolic health (decrease in maternal weight between study inclusion after GDM diagnosis and at 1 yr postpartum) and 2) their mental health (decrease in maternal symptoms of depression during the same time period).

Secondary objective of MySweetHeart Trial:

To test the effect of a multidimensional interdisciplinary lifestyle and psychosocial intervention to improve other cardio-metabolic and mental health markers in women with GDM and their offspring.

MySweetHeart trial is linked to MySweetHeart Cohort, an observational cohort study that assesses the effect of GDM on offspring cardiovascular health early in life. The principal investigators of the cohort are Nicole Sekarski and Arnaud Chiolero (University Hospital Lausanne, Switzerland). Their primary objective is to assess the effect of GDM on the surrogate markers of cardiovascular disease (CVD) at birth (left ventricular mass index and subclinical atherosclerosis) and the secondary objective is to assess the effect of GDM on the cardiovascular structure and function during the fetal period and neonatal adverse cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Women and their partners aged 18 yrs or older, with GDM at 24-32 weeks of gestation, and understanding French or English.

Exclusion Criteria:

* Women on strict bed-rest, with pre-existing diabetes or known severe mental disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
maternal weight measured on calibrated scale | study inclusion after GDM diagnosis and 1 year postpartum
  decrease in maternal weight between study inclusion after GDM diagnosis and 1 year postpartum
Self-reported symptoms of depression (mother) measured by Edinburgh Postnatal Depression Scale | study inclusion after GDM diagnosis and 1 year postpartum
  decrease in maternal symptoms of depression between study inclusion after GDM diagnosis and 1 year postpartum

SECONDARY OUTCOMES:
Body composition (mother and infant) measured by bioelectrical impedance analysis | study inclusion after GDM diagnosis (mother), 6-8 weeks postpartum (mother), 1 year postpartum (infant)
Skinfolds (mother and infant) measured by calipers | study inclusion after GDM diagnosis (mother), 6-8 weeks postpartum (mother), 1 year postpartum (infant)
Total and regional fat mass measured by Dual-Energy X-Ray absorptiometry (mother) | 1 year postpartum
Self-reported food intake (mother) measured by Food Frequency Questionnaire | study inclusion after GDM diagnosis, 1 year postpartum
Self-reported eating behavior (mother) measured by French Intuitive Eating Scale | study inclusion after GDM diagnosis, 1 year postpartum
Self-reported breastfeeding (mother) measured by questionnaire | 6-8- weeks postpartum, 1 year postpartum
Self-reported feeding to soothe (mother) measured by Food to Soothe Questionnaire | 1 year postpartum
Self-reported recognition of hunger/satiety cues (mother) measured by Infant Feeding Style Questionnaire | 1 year postpartum
Physical activity (mother) measured by Accelerometer | study inclusion after GDM diagnosis, 1 year postpartum
Aerobic fitness (mother) measured by Chester Step Test | study inclusion after GDM diagnosis, 1 year postpartum
Grip strength (mother) measured by Jamar dynamometer | study inclusion after GDM diagnosis, 1 year postpartum
Self-reported anxiety (mother) measured by Hospital Anxiety and Depression Scale | study inclusion after GDM diagnosis, 1 year postpartum
Self-reported well-being (mother) measured by WHO Well-being Index | study inclusion after GDM diagnosis, 33-38 weeks GA, 6-8 weeks postpartum,1 year postpartum
Self-reported social support (mother) measured by Medical Outcomes Study Social Support Survey-short form | study inclusion after GDM diagnosis, 1 year postpartum
Weight (infant) measured on calibrated scale | 6-8 weeks postpartum, 1 year postpartum
Laboratory variables (mother): Lipid levels | study inclusion after GDM diagnosis, 6-8 weeks postpartum, 1 year postpartum
Cardiometabolic laboratory variables (mother), HDL cholesterol, LDL cholesterol, total cholesterol, triglycerides, HbA1C, insulin, glucose, indices of insulin resistance and insulin secretion, gamma-GT, B12 vitamin, ferritine, and miRNA | study inclusion after GDM diagnosis, 6-8 weeks postpartum, 1 year postpartum
  Fasting laboratory at inclusion and in addition 75 g oral glucose tolerance test at 6-8 weeks postpartum and 1 year postpartum
Cord blood sample at the time of delivery for lipid levels | At delivery
Cord blood sample at the time of delivery for glucose control | At delivery
Cord blood sample at the time of delivery for insulin indices | At delivery
Cord blood sample at the time of delivery for Ferritin and Vitamin B12 | At delivery
Cord blood sample at the time of delivery for miRNA | At delivery
Laboratory variables (mother): insulin, glucose, indices of insulin resistance and insulin secretion, | study inclusion after GDM diagnosis, 6-8 weeks postpartum, 1 year postpartum
  Fasting laboratory at inclusion and in addition 75 g oral glucose tolerance test at 6-8 weeks postpartum and 1 year postpartum
Laboratory (mother): gamma-GT, B12 vitamin, ferritine | study inclusion after GDM diagnosis, 6-8 weeks postpartum, 1 year postpartum
Laboratory (mother): miRNA | study inclusion after GDM diagnosis, 6-8 weeks postpartum, 1 year postpartum

OTHER OUTCOMES:
Self-reported sleep quality and quantity (mother) measured by Pittsburgh Sleep Quality Index | study inclusion after GDM diagnosis
Self-reported parenting stress (mother) measured by Parenting Stress Scale-short form | 1 year postpartum
Sleep quality and quantity of the infant measured by maternal self-report (Brief Infant Sleep Questionnaire) | 1 year postpartum
Weight of partner measured on calibrated scale | study inclusion after GDM diagnosis, 1 year postpartum
Self-reported eating behavior (partner) measured by French Intuitive Eating Scale | study inclusion after GDM diagnosis, 1 year postpartum
Self-reported well-being (partner) measured by WHO Well-being Index | study inclusion after GDM diagnosis, 1 year postpartum
Self-reported symptoms of depression (partner) measured by Edinburgh Postnatal Depression Scale | study inclusion after GDM diagnosis, 1 year postpartum
Self-reported anxiety (partner) measured by Hospital Anxiety and Depression Scale | study inclusion after GDM diagnosis, 1 year postpartum
Self-reported social support (partner) measured by Medical Outcomes Study Social Support Survey-short form | study inclusion after GDM diagnosis, 1 year postpartum
Self-reported parenting stress (partner) measured by Parenting Stress Scale-short form | 1 year postpartum
Self-reported life events (mother, partner) measured by Life Events Questionnaire | study inclusion after GDM diagnosis, 1 year postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Jardena Puder, MD, Principal Investigator — University of Lausanne Hospitals; Antje Horsch, DClinPsych, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- University Hospital Lausanne, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Quansah DY, Gilbert L, Arhab A, Gonzalez-Rodriguez E, Hans D, Gross J, Lanzi S, Stuijfzand B, Lacroix A, Horsch A, Puder JJ. Effect of a prepartum and postpartum, complex interdisciplinary lifestyle and psychosocial intervention on metabolic and mental health outcomes in women with gestational diabetes mellitus (the MySweetheart trial): randomised, single centred, blinded, controlled trial. BMJ Med. 2024 Feb 7;3(1):e000588. doi: 10.1136/bmjmed-2023-000588. eCollection 2024. PMID 38348309
- [Derived] Gilbert L, Quansah DY, Arhab A, Schenk S, Gross J, Lanzi S, Stuijfzand B, Lacroix A, Horsch A, Puder JJ; MySweetheart Research group. Effect of the MySweetheart randomized controlled trial on birth, anthropometric and psychobehavioral outcomes in offspring of women with GDM. Front Endocrinol (Lausanne). 2023 Jun 7;14:1148426. doi: 10.3389/fendo.2023.1148426. eCollection 2023. PMID 37351105
- [Derived] Horsch A, Gilbert L, Lanzi S, Gross J, Kayser B, Vial Y, Simeoni U, Hans D, Berney A, Scholz U, Barakat R, Puder JJ; MySweetHeart Research Group. Improving cardiometabolic and mental health in women with gestational diabetes mellitus and their offspring: study protocol for MySweetHeart Trial, a randomised controlled trial. BMJ Open. 2018 Feb 27;8(2):e020462. doi: 10.1136/bmjopen-2017-020462. PMID 29487077
- [Derived] Di Bernardo S, Mivelaz Y, Epure AM, Vial Y, Simeoni U, Bovet P, Estoppey Younes S, Chiolero A, Sekarski N; MySweetHeart Research Group. Assessing the consequences of gestational diabetes mellitus on offspring's cardiovascular health: MySweetHeart Cohort study protocol, Switzerland. BMJ Open. 2017 Nov 14;7(11):e016972. doi: 10.1136/bmjopen-2017-016972. PMID 29138200